CLINICAL TRIAL: NCT01386294
Title: A Phase III, Multi-Centre, Randomized Controlled Trial to Assess the Safety and Effectiveness of the Vaginal Microbicide 1% Tenofovir Gel in the Prevention of Human Immunodeficiency Virus Type 1 Infection in Women, and to Examine Effects of the Microbicide on the Incidence of Herpes Simplex Virus Type 2 Infection
Brief Title: Safety and Effectiveness of Tenofovir Gel in the Prevention of Human Immunodeficiency Virus (HIV-1) Infection in Women and the Effects of Tenofovir Gel on the Incidence of Herpes Simplex Virus (HSV-2) Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: Follow-on African Consortium for Tenofovir Studies (FACTS) (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FACTS 001
Record Dates: First submitted 2011-06-28; First posted 2011-07-01 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: HIV Prevention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tenofovir 1% vaginal gel (Experimental): Participants will be required to insert a single dose of assigned gel intravaginally up to 12 hours before coitus and a second dose within 12 hours after coitus but no more than 2 applications within a 24 hour period.
  Interventions: Drug: Tenofovir gel
- Universal placebo gel (Placebo Comparator): Participants will be required to insert a single dose of assigned gel intravaginally up to 12 hours before coitus and a second dose within 12 hours after coitus but no more than 2 applications within a 24 hour period.
  Interventions: Drug: Universal placebo gel

INTERVENTIONS:
Drug: Tenofovir gel — Tenofovir gel is a clear, transparent, viscous gel at concentrations of 1% formulated in purified water with edentate disodium, citric acid, glycerin, methylparaben, propylparaben, HEC, and pH adjusted to 4-5. Tenofovir gel will be supplies in a 4 ml single use applicator containing approximately 4 grams of gel, equivalent to approximately 40mg of tenofovir.
  Arms: Tenofovir 1% vaginal gel
Drug: Universal placebo gel — The placebo gel is an inert gel containing HEC as the gelling agent, purified water, sodium chloride, sorbic acid and sodium hydroxide. Each applicator contains approximately 4ml of placebo gel
  Arms: Universal placebo gel

SUMMARY:
The purpose of the study is to assess the safety and effectiveness of intravaginal 1% tenofovir gel in preventing Human Immunodeficiency Virus (HIV-1) infection and Herpes Simplex Virus (HSV-2) infection in sexually active women.

DETAILED DESCRIPTION:
This is a phase III, multicenter trial to assess the safety and effectiveness of 1% tenofovir gel, administered vaginally by approximately 2900 sexually active women at high risk for sexually transmitted HIV. Approximately 2600 women aged 18-30 years old will be enrolled to achieve the required number of endpoints to show an effect on HIV-1 infection, while up to 300 additional women aged 31-40 years old will be enrolled to collect more safety information in this age group.

This is an event driven study that plans to randomize seronegative women. Participants will be randomized to a 1:1 ratio to receive 1% tenofovir gel or placebo gel. Each will be asked to insert a dose of the assigned study product within 12 hours prior to a coital event and another dose as soon as possible within 12 hours after a coital event. Participants will be advised to use only two doses of gel in a 24 hour period.

All women will be evaluated for the rates of adverse events and the rate of HIV seroconversion. In addition, the study will evaluate several secondary endpoints that bear directly on potential risks and benefits of vaginal tenofovir gel use.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed age 18-40 years (inclusive)
* Able and willing to provide written informed consent
* Able and willing to provide adequate locator information for study retention and safety purposes
* Sexually active, defined as having had vaginal intercourse at least twice in the past 30 days prior to screening
* HIV negative on two rapid tests performed by study staff within 30 days of enrolment (see algorithm in Appendix 3).
* No evidence of glycosuria
* No evidence of proteinuria greater than trace*
* No history of pathological bone fractures
* Have a negative pregnancy test
* Women currently breastfeeding may be enrolled in the study
* Agree to use a study-approved effective non-barrier form of contraception
* Agree to adhere to study visits and procedures
* Willing to use study gel as advised
* Not using or taking any of the following groups of medications:

  * Nephrotoxic agents
  * Drugs that slow renal excretion
  * Immune system modulators
  * Other antiretrovirals

Exclusion Criteria:

* History of adverse reaction to latex.
* Plans any of the following during the study period

  * To travel away from the study site for more than 30 consecutive days.
  * To relocate away from the study site.
  * To become pregnant.
  * To enrol in any other study of an investigational product or behaviour modification related to HIV prevention.
* If in the opinion of the examining clinician, is not sexually active
* Inadequate renal function (serum creatinine greater than 1.5mg/dl and creatinine clearance less than 50ml/min, as estimated using the method of Cockcroft and Gault96 )
* Grade 3 and above ALT and AST at screening or any clinical sign of liver disease ( e.g. ascites, hepatomegaly, jaundice)
* Abnormal serum phosphate levels (Grade 3 and above)
* Has a clinically apparent finding on speculum pelvic examination (observed by study staff) involving deep epithelial disruption. Otherwise eligible participants with speculum pelvic examination findings involving deep epithelial disruption may proceed with enrolment after the findings have resolved and the inclusion/exclusion are met.
* Received previously or receiving an experimental HIV vaccine
* Currently participating in another HIV prevention intervention study or participation in any other clinical trial with a biomedical intervention in the last six months
* Has current STI symptoms and/or other reproductive tract infection requiring treatment, as assessed by study staff. Otherwise eligible participants diagnosed during screening with infection(s) requiring treatment may be enrolled provided that treatment has been completed.
* Any clinical evidence of untreated cervical abnormalities
* Has any other condition that, based on the opinion of the Investigator or designee, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2059 (Actual)
Dates: Start 2011-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Effectiveness | 30 months
  Incidence of HIV-1 infection: HIV incidence will be determine by detection of HIV antibodies using two HIV rapid tests (of which one will be FDA approved) according to algorithm in protocol. One of the rapid tests will detect both HIV-1 and HIV-2; the other will be specific for HIV-1. All endpoints will be reviewed by an expert committee (the Endpoint Adjudication Committee). In carrying out this review, the Committee will use guidelines prepared by the protocol committee for this purpose and recorded in the Manual of Procedures
Safety | 30 months
  Grade 2, 3, and 4 clinical and laboratory adverse events as defined by the DAIDS toxicity table

SECONDARY OUTCOMES:
Incidence of HSV-2 infection | 30 months
  HSV-2 status will be established at enrollment according to a testing algorithm in the protocol. At product discontinuation samples of all those that were HSV-2 seronegative at enrollment will be tested. To identify and confirm incident HSV-2 infections and the timing of these infections, blood samples that were stored will be tested to determine the earliest equivocal or positive result. These samples will be then be tested by HSV Western blot. Samples positive on HSV Western blot will be deemed to be incident HSV-2 infections.
Pregnancy | 30 months
  Incidence of pregnancy loss, prematurity, low birth weight, and major and minor congenital anomalies will be determined
Gel and condom use | 30 months
HIV-1 incidence after product withdrawal | 3 months after product withdrawal
  HIV testing will be conducted 3 months after product discontinuation and if HIV positive, the last stored sample will be tested to ascertain timing of infection and viral tenofovir resistance testing will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Helen Rees, Prof, Study Chair — University of Witwatersrand, South Africa
Locations (9):
- South Africa (9):
  - MatCH Edendale Research Center, Pietermaritzburg, KwaZulu-Natal
  - Desmond Tutu HIV Centre / University of Cape Town, Cape Town
  - Perinatal HIV Research Unit / University of the Witwatersrand, Diepkloof
  - Wits Reproductive Health and HIV Institute / University of the Witwatersrand, Hillbrow
  - Qhakaza Mbokodo Research Clinic, Ladysmith
  - Medunsa Clinical Research Unit / Ga-Ra, Pretoria
  - The Aurum Institute (Rustenburg), Rustenburg
  - Setshaba Research Centre, Soshanguve
  - The Aurum Institute, Tembisa Hospital, Tembisa

REFERENCES:
- [Derived] Delany-Moretlwe S, Lombard C, Baron D, Bekker LG, Nkala B, Ahmed K, Sebe M, Brumskine W, Nchabeleng M, Palanee-Philips T, Ntshangase J, Sibiya S, Smith E, Panchia R, Myer L, Schwartz JL, Marzinke M, Morris L, Brown ER, Doncel GF, Gray G, Rees H. Tenofovir 1% vaginal gel for prevention of HIV-1 infection in women in South Africa (FACTS-001): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2018 Nov;18(11):1241-1250. doi: 10.1016/S1473-3099(18)30428-6. Epub 2018 Oct 24. PMID 30507409